CLINICAL TRIAL: NCT04133831
Title: Don't Throw Your Heart Away: Layperson Study 1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carnegie Mellon University (Other)
Responsible Party: Principal Investigator, Gretchen Chapman, Professor, Carnegie Mellon University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Health Services Research
Other Study IDs: 1 F30 HL152526-01-A; 20PRE35120492 (Other Grant/Funding Number: American Heart Association); 1F30HL152526-01 (NIH)
Record Dates: First submitted 2019-10-18; First posted 2019-10-21 (Actual); Results first posted 2024-10-29 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-08

CONDITIONS: Cardiac Transplant Disorder
Keywords: Heart Transplant; Transplant Survival; Applied Ethics; Decision Psychology; Human Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Condition 1: Combined only (No Intervention): Participants randomized to baseline (control) arm Condition 1 will view only combined transplant survival outcome information (e.g. transplant survival rate not stratified by number and quality of donor hearts accepted at each center) when making a choice between the two hospitals.
- Condition 2: Combined plus Total (Experimental): Participants randomized to Condition 2 will view combined transplant survival and total survival outcome information when making a choice between the two hospitals.
  Interventions: Other: Total Survival
- Condition 3: Stratified only (Experimental): Participants randomized to Condition 3 will view only stratified transplant survival outcome information when making a choice between the two hospitals.
  Interventions: Other: Stratified Transplant Survival
- Condition 4: Stratified plus Total (Experimental): Participants randomized to Condition 4 will view stratified transplant survival and total survival outcome information when making a choice between the two hospitals.
  Interventions: Other: Total Survival; Other: Stratified Transplant Survival
- Condition 5: Total only (Experimental): Participants randomized to Condition 5 will view only total survival outcome information when making a choice between the two hospitals.
  Interventions: Other: Total Survival

INTERVENTIONS:
Other: Total Survival — The overall or "total" survival rate at each center is displayed in the table of outcome statistics.
  Total survival is computed from survival rates of both transplant and waitlist patients: [(number of patients surviving after transplant at end of year + number of patients alive on waitlist at end of year)] / [number of patients alive on waitlist at start of year].
  Arms: Condition 2: Combined plus Total; Condition 4: Stratified plus Total; Condition 5: Total only
Other: Stratified Transplant Survival — The transplant survival rate in the table of outcome statistics is stratified into two groups: (i) patients who received excellent donor organs and (ii) patients who received less than optimal donor organs.
  Stratified transplant survival is computed from survival rates of transplant patients who received each quality category of organ.
  excellent transplant survival = [number of patients surviving after transplant with excellent organ]/[number of patients for whom excellent organ was accepted for transplant] marginal transplant survival = [number of patients surviving after transplant with marginal organ]/[number of patients for whom marginal organ was accepted for transplant]
  Arms: Condition 3: Stratified only; Condition 4: Stratified plus Total

SUMMARY:
Publicly available outcome assessments for transplant programs do not make salient that some programs tend to reject many of the hearts they are offered, whereas other programs accept a broader range of donor offers. The investigators use empirical studies to test whether transplant center performance data (i.e. transplant and waitlist outcome statistics) that reflect center donor acceptance rates influence laypersons to evaluate centers with high organ decline rates less favorably than centers with low organ decline rates. 1000 lay participants will be recruited from Amazon Mechanical Turk and randomized to one of five different information presentation conditions. Participants will be given an introduction to the donor organ match process, then asked to view the table of transplant outcomes corresponding to the condition they were randomized to. Each participant is asked to choose between two hospitals: one hospital with an non-selective, "accepting" strategy (takes all donor heart offers), and one hospital with a more selective, "cherrypicking" strategy (tends to reject donor offers that are less than "excellent" quality).

DETAILED DESCRIPTION:
Publicly available outcome assessments for transplant programs do not make salient that some programs tend to reject many of the hearts they are offered, whereas other programs accept a broader range of donor offers. The investigators use empirical studies to test whether transplant center performance data (i.e. transplant and waitlist outcome statistics) that reflect center donor acceptance rates influence laypersons to evaluate centers with high organ decline rates less favorably than centers with low organ decline rates. 1000 lay participants will be recruited from Amazon Mechanical Turk and randomized to one of five different information presentation conditions:

1. Condition 1 ("baseline" condition): view only combined transplant survival (e.g. transplant survival rate not stratified by number and quality of donor hearts accepted at each center)
2. Condition 2: view combined transplant survival + total survival (e.g. overall survival rate at each center, computed from survival rates of both transplant and waitlist patients)
3. Condition 3: view only stratified transplant survival (e.g. transplant survival rate stratified into patients who received excellent donor organs and patients who received less than optimal donor organs)
4. Condition 4: view stratified transplant survival + total survival
5. Condition 5: view only total survival

Participants will be given an introduction to the donor organ match process, then asked to view the table of transplant outcomes corresponding to the condition they were randomized to. Each participant is asked to choose between two hospitals: one hospital with an non-selective, "accepting" strategy (takes all donor heart offers), and one hospital with a more selective, "cherrypicking" strategy (tends to reject donor offers that are less than "excellent" quality). In order to identify the decision process that underlies this choice pattern, the investigators will examine a putative mediator. Specifically, participants will be asked to rate the extent to which they considered patients' chances of getting an excellent heart, avoiding a less-than-optimal heart, and getting any type of heart when making their choice between the two hospitals.

ELIGIBILITY:
Inclusion Criteria:

Participants who are already qualified mTurk workers with Worker Accounts meeting the above criteria will be asked to participate if they confirm the following inclusion criteria in the consent form.

1. 18 years of age or older
2. must read and understand the information in the consent form
3. must want to participate in the research and continue with the survey
4. must live in United States

Exclusion Criteria:

1. Participants on mTurk will not be allowed to participate if they fail to pass the initial "bot screening", a multiple-choice question that asks, "What phone number should you dial when there is an emergency?" The obvious correct response in this screening question is "911", so participants who select one of the incorrect responses (i.e. "1-800-ANTIBOT", "1-877-MTURKER", "123") are filtered out and not allowed to complete the survey.
2. Participants on mTurk will be allowed to participate, but excluded from data analysis, if they submit a nonsense response to the free-response question which reads, "In your own words, why do you think patients should choose the hospital you picked?" This question takes place after the participant has viewed the choice stimuli and selected their response. If participants input nonsense in the text response box, they will be permitted to complete the survey and paid, but filtered out from the data analysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1019 (Actual)
Dates: Start 2019-11-15 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alison E Butler, BS, Principal Investigator — Carnegie Mellon University
Locations (1):
- Carnegie Mellon University, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
The PI will make all of the raw IPD files - together with statistical analysis protocol descriptions and information for proper analysis available for download a minimum of 1 year, and a maximum of 3 years, after publication of the corresponding manuscripts. All human subjects data are anonymized immediately when they are initially written from the online survey platform to the server, and thus participant confidentiality will not be compromised by this plan for data sharing.
  All hypotheses, methods, and planned analyses for the applicant's studies will be pre-registered on ClinicalTrials.gov and Open Science Framework.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: All of the raw files, statistical analysis protocol descriptions, and information for proper analysis will be available for download a minimum of 1 year, and a maximum of 3 years, after publication of the corresponding manuscripts.
URL: https://osf.io/9fsb3/

RESULTS

PARTICIPANT FLOW:
Groups:
- Condition 2: Combined Plus Total: Participants randomized to Condition 2 will view combined transplant survival and total survival outcome information when making a choice between the two hospitals.
  Total Survival: The overall or "total" survival rate at each center is displayed in the table of outcome statistics.
  Total survival is computed from survival rates of both transplant and waitlist patients: [(number of patients surviving after transplant at end of year + number of patients alive on waitlist at end of year)] / [number of patients alive on waitlist at start of year].
- Condition 3: Stratified Only: Participants randomized to Condition 3 will view only stratified transplant survival outcome information when making a choice between the two hospitals.
  Stratified Transplant Survival: The transplant survival rate in the table of outcome statistics is stratified into two groups: (i) patients who received excellent donor organs and (ii) patients who received less than optimal donor organs.
  Stratified transplant survival is computed from survival rates of transplant patients who received each quality category of organ.
  excellent transplant survival = [number of patients surviving after transplant with excellent organ]/[number of patients for whom excellent organ was accepted for transplant] marginal transplant survival = [number of patients surviving after transplant with marginal organ]/[number of patients for whom marginal organ was accepted for transplant]
- Condition 4: Stratified Plus Total: Participants randomized to Condition 4 will view stratified transplant survival and total survival outcome information when making a choice between the two hospitals.
  Total Survival: The overall or "total" survival rate at each center is displayed in the table of outcome statistics.
  Total survival is computed from survival rates of both transplant and waitlist patients: [(number of patients surviving after transplant at end of year + number of patients alive on waitlist at end of year)] / [number of patients alive on waitlist at start of year].
  Stratified Transplant Survival: The transplant survival rate in the table of outcome statistics is stratified into two groups: (i) patients who received excellent donor organs and (ii) patients who received less than optimal donor organs.
  Stratified transplant survival is computed from survival rates of transplant patients who received each quality category of organ.
  excellent transplant survival = [number of patients surviving after transplant with excellent organ]/[number of patients for whom excellent organ was accepted for transplant] marginal transplant survival = [number of patients surviving after transplant with marginal organ]/[number of patients for whom marginal organ was accepted for transplant]
- Condition 5: Total Only: Participants randomized to Condition 5 will view only total survival outcome information when making a choice between the two hospitals.
  Total Survival: The overall or "total" survival rate at each center is displayed in the table of outcome statistics.
  Total survival is computed from survival rates of both transplant and waitlist patients: [(number of patients surviving after transplant at end of year + number of patients alive on waitlist at end of year)] / [number of patients alive on waitlist at start of year].
Period: Overall Study
Arm/Group | Condition 1: Combined Only | Condition 2: Combined Plus Total | Condition 3: Stratified Only | Condition 4: Stratified Plus Total | Condition 5: Total Only
Started | 183 | 194 | 192 | 209 | 241
Completed | 183 | 194 | 192 | 209 | 241
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Condition 1: Combined Only | Condition 2: Combined Plus Total | Condition 3: Stratified Only | Condition 4: Stratified Plus Total | Condition 5: Total Only | Total
Number analyzed (Participants) | 183 | 194 | 192 | 209 | 241 | 1019
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 0 | 0 | 0 | 1
  Between 18 and 65 years | 181 | 192 | 190 | 207 | 239 | 1009
  >=65 years | 1 | 2 | 2 | 2 | 2 | 9
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Sex/Gender (customized): Female | 82 | 97 | 87 | 102 | 119 | 487
  Sex/Gender (customized): Male | 97 | 90 | 96 | 106 | 115 | 504
  Sex/Gender (customized): Unknown/Other | 4 | 7 | 9 | 1 | 7 | 28
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 2 | 1 | 0 | 1 | 6
  Asian | 9 | 7 | 10 | 11 | 11 | 48
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 0 | 0 | 0 | 2
  Black or African American | 13 | 10 | 14 | 19 | 16 | 72
  White | 142 | 154 | 141 | 157 | 190 | 784
  More than one race | 6 | 11 | 9 | 10 | 13 | 49
  Unknown or Not Reported | 9 | 10 | 17 | 12 | 10 | 58
Region of Enrollment [Number; unit: participants]
  United States | 183 | 194 | 192 | 209 | 241 | 1019

OUTCOME MEASURES:

1. Primary Outcome: Hospital Choice
Description: The outcome variable will be a measure of binary choice between two hospitals: one with a selective donor-heart acceptance strategy and one with a non-selective donor heart acceptance strategy.
  Participants will respond to the question "Which Hospital is a better choice for patients? Please click on one of the two tables below to indicate which hospital is the better choice." Participants will choose been two outcome tables featuring the selective and non-selective hospital (counterbalanced, such that each of the two choices is equally likely to be presented at top of the choice scenario in each condition). The number of participants that choose each hospital will be the measured outcome variable used in analyses.
Time Frame: 1 day
Measure: Count of Participants; unit: Participants
Arm/Group | Condition 1: Combined Only | Condition 2: Combined Plus Total | Condition 3: Stratified Only | Condition 4: Stratified Plus Total | Condition 5: Total Only
Number analyzed (Participants) | 183 | 194 | 192 | 209 | 241
Participants
  Proportion choosing non-selective center | 64 | 125 | 163 | 192 | 224
  Proportion choosing selective center | 119 | 69 | 29 | 17 | 17

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Condition 1: Combined Only | Condition 2: Combined Plus Total | Condition 3: Stratified Only | Condition 4: Stratified Plus Total | Condition 5: Total Only
All-Cause Mortality (participants affected / at risk) | 0/183 | 0/194 | 0/192 | 0/209 | 0/241
Serious Adverse Events (participants affected / at risk) | 0/183 | 0/194 | 0/192 | 0/209 | 0/241
Other Adverse Events (participants affected / at risk) | 0/183 | 0/194 | 0/192 | 0/209 | 0/241

LIMITATIONS AND CAVEATS:
Selection bias or underrepresentation of certain groups due to online worker platform.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-01-10): https://cdn.clinicaltrials.gov/large-docs/31/NCT04133831/Prot_SAP_000.pdf